CLINICAL TRIAL: NCT04645238
Title: Comparison of the Effects of Static and PNF Hamstring Stretching Exercises in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ilke KARA, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEU-FTR-IK-01
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Hamstring; Stretching
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Static Hamstring Stretching (Active Comparator): Static Hamstring Stretching
  Interventions: Other: Static Stretching
- PNF Stretching (Active Comparator): PNF Hamstring Stretching (Hold-Relax)
  Interventions: Other: PNF Stretching

INTERVENTIONS:
Other: Static Stretching — Static hamstring stretching exercise lasting 30 seconds and 10 repetitions under the supervision of the physiotherapist
  Arms: Static Hamstring Stretching
Other: PNF Stretching — PNF hold-relax stretching technique that consists of 10 seconds isometric contraction, 30 seconds hamstring stretching and 10 repetitions under the supervision of the physiotherapist
  Arms: PNF Stretching

SUMMARY:
The aim of this study is to determine and compare the effects of static and PNF hamstring stretching exercises on joint pain, hamstring flexibility and functional status in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A total of 36 patients between the ages of 40 and 75 who were diagnosed with Kellgren-Lawrence Stage II and III knee OA by the physician were included in the study. Participants were divided into two groups as static stretching group or PNF stretching group. Patients' demographic and clinical information was recorded. Pain intensity was evaluated with visual pain scale, hamstring flexibility with Active Knee Extension Test, functional status with Western Ontario and McMasters University Osteoarthritis Index and Timed Get Up and Go Test. In addition to the standard physiotherapy program, the subjects practiced stretching exercises according to the groups that they've been separated. Evaluations were repeated in the end of the treatment and in the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with knee osteoarthritis severity II, III, or IV according to the Kellgren-Lawrence Classification,
* Individuals with positive active knee extension test,
* Individuals with a body mass index of 30 or less,
* Individuals with a pain severity of at least 3/10 according to the visual pain scale.

Exclusion Criteria:

* Individuals with health problems that prevent them from doing the evaluations and exercises to be used in the study,
* Individuals who exercise regularly for the last six months,
* Individuals with a diagnosis of neurological disease affecting the lower extremity.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test for Hamstring Flexibility | Baseline and post-intervention
  Higher values represent better outcomes.
Active Knee Extension Test for Hamstring Flexibility | Post-intervention and follow-up
  Higher values represent better outcomes.

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain | Baseline and post-intervention
  The scale varies from 0 to 10. Higher values represent worse outcomes.
Visual Analogue Scale for Pain | Post-intervention and follow-up
  The scale varies from 0 to 10. Higher values represent worse outcomes.
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline and post-intervention
  The scale varies from 0 to 96. Higher values represent worse outcomes.
Western Ontario and McMaster Universities Osteoarthritis Index | Post-intervention and follow-up
  The scale varies from 0 to 96. Higher values represent worse outcomes.
The Timed Up & Go Test | Baseline and post-intervention
  Higher values represent worse outcomes.
The Timed Up & Go Test | Post-intervention and follow-up
  Higher values represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Gelecek, Professor, Study Director — Dokuz Eylul University
Locations (1):
- Fizyotem Medical Center, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid DA, McNair PJ. Effects of an acute hamstring stretch in people with and without osteoarthritis of the knee. Physiotherapy. 2010 Mar;96(1):14-21. doi: 10.1016/j.physio.2009.06.010. Epub 2009 Sep 4. PMID 20113758
- [Background] Hortobagyi T, Westerkamp L, Beam S, Moody J, Garry J, Holbert D, DeVita P. Altered hamstring-quadriceps muscle balance in patients with knee osteoarthritis. Clin Biomech (Bristol). 2005 Jan;20(1):97-104. doi: 10.1016/j.clinbiomech.2004.08.004. PMID 15567543
- [Background] Krishnasamy P, Hall M, Robbins SR. The role of skeletal muscle in the pathophysiology and management of knee osteoarthritis. Rheumatology (Oxford). 2018 May 1;57(suppl_4):iv22-iv33. doi: 10.1093/rheumatology/kex515. PMID 29351644
- [Background] Rutherford DJ, Hubley-Kozey CL, Stanish WD. Changes in knee joint muscle activation patterns during walking associated with increased structural severity in knee osteoarthritis. J Electromyogr Kinesiol. 2013 Jun;23(3):704-11. doi: 10.1016/j.jelekin.2013.01.003. Epub 2013 Jan 26. PMID 23357547
- [Background] Lempke L, Wilkinson R, Murray C, Stanek J. The Effectiveness of PNF Versus Static Stretching on Increasing Hip-Flexion Range of Motion. J Sport Rehabil. 2018 May 1;27(3):289-294. doi: 10.1123/jsr.2016-0098. Epub 2018 May 22. PMID 28182516
- [Background] Lim KI, Nam HC, Jung KS. Effects on hamstring muscle extensibility, muscle activity, and balance of different stretching techniques. J Phys Ther Sci. 2014 Feb;26(2):209-13. doi: 10.1589/jpts.26.209. Epub 2014 Feb 28. PMID 24648633
- [Background] Hill KJ, Robinson KP, Cuchna JW, Hoch MC. Immediate Effects of Proprioceptive Neuromuscular Facilitation Stretching Programs Compared With Passive Stretching Programs for Hamstring Flexibility: A Critically Appraised Topic. J Sport Rehabil. 2017 Nov;26(6):567-572. doi: 10.1123/jsr.2016-0003. Epub 2016 Aug 24. PMID 27632820
- [Background] Maddigan ME, Peach AA, Behm DG. A comparison of assisted and unassisted proprioceptive neuromuscular facilitation techniques and static stretching. J Strength Cond Res. 2012 May;26(5):1238-44. doi: 10.1519/JSC.0b013e3182510611. PMID 22395273
- [Background] Fasen JM, O'Connor AM, Schwartz SL, Watson JO, Plastaras CT, Garvan CW, Bulcao C, Johnson SC, Akuthota V. A randomized controlled trial of hamstring stretching: comparison of four techniques. J Strength Cond Res. 2009 Mar;23(2):660-7. doi: 10.1519/JSC.0b013e318198fbd1. PMID 19204565
- [Background] Yildirim MS, Ozyurek S, Tosun O, Uzer S, Gelecek N. Comparison of effects of static, proprioceptive neuromuscular facilitation and Mulligan stretching on hip flexion range of motion: a randomized controlled trial. Biol Sport. 2016 Mar;33(1):89-94. doi: 10.5604/20831862.1194126. Epub 2016 Feb 8. PMID 26929476
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Song Q, Shen P, Mao M, Sun W, Zhang C, Li L. Proprioceptive neuromuscular facilitation improves pain and descending mechanics among elderly with knee osteoarthritis. Scand J Med Sci Sports. 2020 Sep;30(9):1655-1663. doi: 10.1111/sms.13709. Epub 2020 Jun 1. PMID 32407583